CLINICAL TRIAL: NCT01942200
Title: Open, Multicenter Observational Study of Oxaliplatin Utilized in Combination Therapy for Adjuvant Treatment of Colon Carcinoma of Stage III After Complete Removal of the Primary Tumor and for Treatment of Metastasizing Colorectal Carcinoma.
Brief Title: A Non Interventional Study With Oxaliplatin Onkovis (Oxaliplatin) Utilized for the Treatment of Cancer
Status: Completed | Type: Observational
Sponsor: Onkovis GmbH (Industry)
Collaborators: AKP Freiburg GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: ONKOOXA01
Record Dates: First submitted 2013-09-10; First posted 2013-09-13 (Estimated); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Carcinoma
Keywords: carcinoma; colon cancer; colorectal cancer; ambulant chemotherapy; treatment cycles; Oxaliplatin; Oxaliplatin onkovis; Quantity of Oxaliplatin; Packaging Sizes
MeSH Terms: conditions — Carcinoma; Colonic Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Carcinoma, Oxaliplatin onkovis (Oxaliplatin): Treatment in combination therapy for adjuvant treatment of colon carcinoma of stage III (Dukes C) after complete removal of the primary tumor, as well as for treatment of metastasizing colorectal carcinoma.

SUMMARY:
The main purpose of this observational study with Oxaliplatin onkovis is to determine the number of treatment cycles and the quantity of Oxaliplatin onkovis needed for this purpose under the special circumstances of ambulant chemotherapy.

Onkovis aims to contribute to an economical utilization of the chemotherapeutics. This includes provision of appropriate packaging sizes to decrease the excess quantity to be discarded, and thus also follows this objective.

Secondary objective is the assessment of the side effects of Oxaliplatin onkovis. To this end, data regarding co-medication and adverse events are also collected.

ELIGIBILITY:
Inclusion Criteria:

* Indication for Oxaliplatin according to the Summary of Product Characteristics (SmPC) and treating physician

Exclusion Criteria:

* According to the Oxaliplatin SmPC

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated in practices, clinics, hospitals
Sampling Method: Probability Sample
Enrollment: 383 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
The Quantity of Oxaliplatin onkovis needed per treatment cycle | up to 24 weeks
  Determine the quantity of Oxaliplatin onkovis needed per treatment cycle

SECONDARY OUTCOMES:
Adverse events during and after treatment | up to 24 weeks
  The number and type of adverse events during and after the intra-venous application of Oxaliplatin will be assessed and documented.

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Practice, Elstra
  - Practice, Leipzig
  - Practice, Naunhof